CLINICAL TRIAL: NCT03534323
Title: A Phase I/II Study of Duvelisib and Venetoclax in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma or Patients With Richter's Syndrome
Brief Title: Duvelisib and Venetoclax in Relapsed or Refractory CLL or SLL or RS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Secura Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-089
Record Dates: First submitted 2018-05-02; First posted 2018-05-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia; Richter Syndrome
Keywords: chronic lymphocytic leukemia (CLL); Richter's Syndrome; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib +Venetoclax, (Experimental): Duvelisib will be given alone for the first seven days. On day 8 Venetoclax will be added.
  * Duvelisib will be administered orally twice daily
  * Venetoclax will be administered orally daily
  * All patients will be admitted for administration of the initial dose of venetoclax at each dose escalation
  Interventions: Drug: Duvelisib; Drug: Venetoclax

INTERVENTIONS:
Drug: Duvelisib — This drug is designed to stop cancer growth by blocking a protein called phosphatidylinositide 3-kinase (PI3K), which is important for the survival of CLL cells.
  Other Names: IPI-145
Drug: Venetoclax — Venetoclax targets a protein called BCL-2, which helps cancer cells survive.
  Other Names: Venclexta

SUMMARY:
This research study is assessing a new drug, duvelisib, in combination with a drug that is already FDA approved, venetoclax, as a possible treatment for participants with CLL or those with Richter's Syndrome

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational drugs and also tries to define the appropriate dose of the investigational drugs to use for further studies. "Investigational" means that the drugs are being studied together for the first time.

This phase I study tests the safety of the drug duvelisib when used in combination with the drug venetoclax. Duvelisib is still being studied, but the FDA (the U.S. Food and Drug Administration) has approved the use of Duvelisib in patients with CLL/SLL with relapsed or refractory CLL after having received 2 or more prior therapies.

Duvelisib is a drug that is given in capsule form and taken by mouth. This drug is designed to stop cancer growth by blocking a protein called phosphatidylinositide 3-kinase (PI3K), which is important for the survival of CLL cells. In laboratory studies and in other clinical trials that included participants with CLL, duvelisib was effective at killing CLL cells.

Venetoclax is a tablet that is taken by mouth. Venetoclax targets a protein called BCL-2, which helps cancer cells survive. Venetoclax is an effective treatment for many participants with CLL who do not respond to chemotherapy or other approved drugs or who have relapsed after prior therapy.Venetoclax is FDA approved for participants with CLL who have never had therapy before or whose CLL has worsened after prior therapy.

In the phase I portion of this study, the investigators are looking to determine the dose of venetoclax that is safe to give with duvelisib and to see what the side effects are of this combination.

In the phase II portion of this study, we are looking to determine how effective thecombination of duvelisib and venetoclax is for patients with CLL or Richter's Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma requiring therapy, as per IW-CLL 2008 criteria OR Biopsy proven transformation to diffuse large B cell lymphoma (DLBCL), consistent with Richter's Syndrome
* Disease that has progressed during or relapsed after at least one previous CLL/SLL therapy - If Richter's Syndrome, this criterion is not applicable
* Age greater to or equal to 18 years
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of CLL confirmed on biopsy:

  * Absolute neutrophil count ≥500 cells/mm3 (0.5 x 109/L). Growth factor is allowed in order to achieve this
  * Platelet count ≥25,000 cells/mm3 (25 x 109/L) independent of transfusion within 7 days of screening
* Adequate hepatic function defined as:

  --Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN), bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Adequate renal function as defined as:

  --Serum creatinine ≤1.5 times the upper limit of normal or creatinine clearance ≥ 50 mL/min using a 24-hour urine collection
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method or abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Previous treatment with venetoclax or duvelisib
* Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, surgery within 2 weeks of Cycle 1/Day 1 with the following exceptions:

  * For patients on targeted therapies, a washout of least five half lives is required
  * Patients who experience clinical deterioration may start therapy after a shorter washout period with prior approval by the PI
  * Corticosteroid therapy (prednisone or equivalent <20 mg daily) is allowed
* Confirmed central nervous system involvement
* Allogeneic hematologic stem cell transplant within 6 months of starting study treatment or active graft vs. host disease (GVHD) requiring treatment or prophylaxis
* History of active malignancy requiring therapy with the exception of hormonal therapy
* Any active systemic infection requiring IV antibiotics or uncontrolled, active infections
* Known history of human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV)
* Major surgery within 4 weeks of first dose of study drug
* Currently active gastrointestinal disease, including colitis, inflammatory bowel disease and diarrhea requiring therapy
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Use of Coumadin for anticoagulation (other anticoagulants permitted)
* Lactating or pregnant
* Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A (see Appendix D) . The concomitant use of drugs or foods that are strong or moderate inhibitors or inducers of CYP3A are not allowed beginning 1 week prior to the first dose of duvelisib.
* Patients with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not included on the list of prohibited medications
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction resulting in malabsorption or chronic diarrhea
* Active abuse of alcohol
* History of chronic liver disease or veno-occlusive disease/sinusoidal obstruction syndrome
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* Known hypersensitivity to duvelisib and/or its excipients
* History of tuberculosis treatment within the 2 years prior to initiation of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Venetoclax When Administered with Duvelisib | Up to 7 weeks
  As assessed by protocol-specified DLT criteria (phase I)
Rate of complete remission | 2 years
  By IW-CLL criteria (phase II)

SECONDARY OUTCOMES:
Cmax | Up to 7 weeks
  Cmax
Half-life | Up to 7 weeks
  Half-life
Volume of Distribution | Up to 7 weeks
  Volume of Distribution
Objective response rate | 2 years
  By IW-CLL Criteria
Duration of response | 2 years
  By IW-CLL Criteria
Progression free survival | 2 years
  By IW-CLL Criteria
Rate of minimal residual disease negativity | 2 years
  By IW-CLL Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Davids, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - University of Miami- Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northern Light Eastern Maine Medical Center, Brewer, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts

IPD SHARING:
Plan to Share IPD: No